CLINICAL TRIAL: NCT05559099
Title: A Randomized, Placebo-controlled, Double-blinded Trial of the Safety and Efficacy of Tecovirimat for the Treatment of Adult and Pediatric Patients With Monkeypox Virus Disease
Brief Title: Tecovirimat for Treatment of Monkeypox Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PALM 007
Record Dates: First submitted 2022-09-23; First posted 2022-09-29 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Monkeypox
Keywords: Monkeypox; MPXV
MeSH Terms: conditions — Mpox, Monkeypox | interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tecovirimat (Experimental): Tecovirimat capsules administered orally to participants for 14 days plus SOC.
  Interventions: Drug: Tecovirimat Oral Capsule
- Placebo (Placebo Comparator): Matching placebo capsules administered orally to participants for 14 days plus SOC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tecovirimat Oral Capsule — 200 mg capsules
  Number of capsules and frequency of dosage will be based on participant weight:
  * ≥120 kg: three capsules three times a day (total daily tecovirimat dose: 1,800 mg)
  * 40 to <120 kg: three capsules twice a day (total daily tecovirimat dose: 1,200 mg)
  * 25 to <40 kg: two capsules twice a day (total daily tecovirimat dose: 800 mg)
  * 13 to <25 kg: one capsule twice a day (total daily tecovirimat dose: 400 mg)
  * 6 to <13 kg: ½ the contents of a capsule twice daily (total daily tecovirimat dose: 200 mg)
  * 3 to <6 kg: ¼ the contents of a capsule twice daily (total daily tecovirimat dose: 100 mg)
  Other Names: TPOXX
  Arms: Tecovirimat
Drug: Placebo — Capsules to match tecovirimat
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if tecovirimat is a safe and effective drug to treat monkeypox (mpox) in combination with standard of care (SOC). Participants will be randomly assigned to receive oral tecovirimat plus SOC or placebo plus SOC for 14 days.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind study to test the antiviral drug tecovirimat for the treatment of adults and children with laboratory-confirmed monkeypox virus (MPXV) disease at participating sites in the Democratic Republic of Congo. Eligible and consented participants will be randomized 1:1 to receive either oral tecovirimat or placebo, each administered in the hospital with standard-of-care (SOC) treatment for 14 days. Participants will be followed for 28 days with an optional visit at Day 59 for long-term assessment.

If a participant reaches full body lesion resolution but subsequently develops at least one new lesion consistent with mpox after discharge but while still enrolled in the study, they will be eligible to make a sick visit and will be offered standard of care for mpox.

ELIGIBILITY:
This study has no age restriction.

Inclusion Criteria:

* Laboratory-confirmed monkeypox virus infection as determined by PCR obtained from blood, oropharynx, or skin lesion within 48 hours of screening
* Monkeypox illness of any duration provided that the patient has at least one active, not yet scabbed, lesion
* Weight ≥3 kg
* Men and non-pregnant women of reproductive potential must agree to use effective means of contraception when engaging in sexual activities that can result in pregnancy, from the time of enrollment through the end of study participation. Acceptable methods of contraception include the following:

  * Hormonal contraception
  * Male or female condom
  * Diaphragm or cervical cap with a spermicide
  * Intrauterine device
* Stated willingness to comply with all study procedures (including required inpatient stay) and availability for the duration of the study
* Ability to provide informed consent personally or by a legally or culturally acceptable representative if the patient is unable to do so

Exclusion Criteria:

* Current or planned use of a meglitinide (repaglinide, nateglinide)
* Planned use of midazolam while on study drug
* Severe anemia, defined as hemoglobin <7 g/dL
* Current or planned use of another investigational drug at any point during study participation
* Patients who, in the judgement of the investigator, will be at significantly increased risk as a result of participation in the study
* Participants who are unable to safely swallow oral medications, such as those who are at risk of aspiration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Muyembe-Tamfum, MD PhD, Principal Investigator — Kinshasa University
Locations (2):
- Democratic Republic of the Congo (2):
  - L'Hôpital Général de Référence de Kole, Kole
  - L'Hôpital Général de Référence de Tunda, Tunda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] PALM007 Writing Group; Ali R, Alonga J, Biampata JL, Kombozi Basika M, Maljkovic Berry I, Bisento N, Blum E, Bonnett T, Cone K, Crozier I, Davey R, Dilu A, Dodd LE, Gulati I, Hruby D, Ibanda A, Isse F, Kasareka SS, Kayembe G, Kojan R, Luzolo EK, Lane HC, Lawanga L, Liesenborghs L, Shosongo Lunghe C, Lula Y, Lusakibanza M, Lutete GT, Mbala-Kingebeni P, Miranda A, Mukadi-Bamuleka D, Mukendi G, Lupola PM, Muyembe-Tamfum JJ, Ndungunu R, Nganga B, Ntamabyaliro N, Nussenblatt V, Omulepu I, Omalokoho Onosomba J, Proschan M, Rubenstein K, Saknite I, Schechner A, Shaw-Saliba K, Sivahera B, Smolskis M, Tillman A, Tkaczyk E, Tshimanga C, Tshiani Mbaya O, Tshomba A, Yemba Unda Tshomba F, Vallee D, Vogel S, Weyers S. Tecovirimat for Clade I MPXV Infection in the Democratic Republic of Congo. N Engl J Med. 2025 Apr 17;392(15):1484-1496. doi: 10.1056/NEJMoa2412439. PMID 40239067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the areas surrounding two sites in rural Democratic Republic of the Congo - Tunda and Kole. Patient recruitment took place from October 2022 through July 9, 2024.
Period: Overall Study
Arm/Group | Tecovirimat | Placebo
Started | 295 | 302
Completed | 289 | 295
Not Completed | 6 | 7
Not completed — Death | 5 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat primary analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecovirimat | Placebo | Total
Number analyzed (Participants) | 295 | 302 | 597
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.4 (13.9) | 15.3 (13.9) | 15.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 151 | 292
  Male | 154 | 151 | 305
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Days since onset of symptoms [Mean (Standard Deviation); unit: Days] — Number of days since patient-reported onset of mpox symptoms
  Days | 5.9 (2.5) | 5.9 (2.8) | 5.9 (2.6)
Less than or equal to 7 days since onset of symptoms [Count of Participants; unit: Participants] — Grouped number of days since patient-reported onset of mpox symptoms
  Participants | 234 | 239 | 473
Greater than 7 days since onset of symptoms [Count of Participants; unit: Participants] — Grouped number of days since patient-reported onset of mpox symptoms
  Participants | 61 | 63 | 124

OUTCOME MEASURES:

1. Primary Outcome: Time to Lesion Resolution
Description: Number of days from randomization to the first day on which all lesions on the total body are scabbed or desquamated or a new layer of epidermis has formed.
Time Frame: Up to day 28
Population: Intention to treat population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 295 | 302
Days | 7 [7 to 8] | 8 [7 to 9]

2. Secondary Outcome: Time to Lesion Resolution for Participants With Symptom Onset Less Than or Equal to 7 Days Before Randomization
Description: Number of days to the first day on which all lesions on the total body are scabbed or desquamated or a new layer of epidermis has formed.
Time Frame: up to day 28
Population: Intention to treat population - participants with symptom onset less than or equal to 7 days before randomization
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 234 | 239
Days | 7 [7 to 8] | 8 [7 to 8]

3. Secondary Outcome: Time to Lesion Resolution for Participants With Symptom Onset Greater Than 7 Days Before Randomization
Description: as for outcome 2
Time Frame: up to day 28
Population: Intention to treat population - participants with symptom onset greater than 7 days before randomization
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 61 | 63
Days | 8 [7 to 10] | 8 [7 to 11]

4. Secondary Outcome: Number and Percentage of Participants With Negative Blood PCR Results
Description: Percentage of participants with negative blood sample MPXV PCR results 14 days post-randomization, out of those positive at baseline
Time Frame: day 14
Population: Intention to treat population - participants with positive MPXV PCR in the blood at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 160 | 162
Participants | 140 | 141

5. Secondary Outcome: Number and Percentage of Participants With Negative Oropharyngeal Swab PCR Results
Description: Number and percentage of participants with negative oropharyngeal swab MPXV PCR results 14 days post-randomization, out of those positive at baseline
Time Frame: day 14
Population: Intention to treat population - participants with positive oropharyngeal swab MPXV PCR results at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 260 | 259
Participants | 144 | 136

6. Secondary Outcome: Number and Percentage of Participants With Negative Lesion Swab PCR Results
Description: Number and and percentage of participants with negative lesion swab MPXV PCR results 14 days post-randomization, of those positive at baseline
Time Frame: day 14
Population: Intention to treat population - participants with positive lesion swab MPXV PCR results at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 280 | 291
Participants | 256 | 259

7. Secondary Outcome: Mortality Within the First 28 Days Post-randomization
Description: Number of deaths post-randomization
Time Frame: up to day 28
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 295 | 302
Participants | 3 | 4

8. Secondary Outcome: Incidence of Non-fatal Serious Adverse Events Requiring Permanent Drug Discontinuation
Description: Number of participants with a non-fatal serious adverse event requiring permanent drug discontinuation through the end of the treatment period (14 days)
Time Frame: Up to day 14
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 295 | 302
Participants | 0 | 2

9. Secondary Outcome: Incidence of Non-fatal Adverse Events Requiring Permanent Drug Discontinuation
Description: Number of participants with a non-fatal adverse event requiring permanent drug discontinuation through the end of the treatment period (14 days)
Time Frame: Up to day 14
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 295 | 302
Participants | 1 | 0

10. Secondary Outcome: Incidence of Adverse Events
Description: Number of participants with an adverse event up to day 28
Time Frame: up to day 28
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 295 | 302
Participants | 196 | 199

11. Secondary Outcome: Incidence of Bacterial Infection Adverse Events
Description: Number of participants with a bacterial infection adverse event up to day 28
Time Frame: up to day 28
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Tecovirimat | Placebo
Number analyzed (Participants) | 295 | 302
Participants | 23 | 27

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 58 days
Description: All adverse events were documented and recorded and all grade 3 and above adverse events were reported to a study pharmacovigilance committee from the time informed consent was obtained through the end of subject participation in the study. Where possible, adverse events were graded according to the "Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Laboratory values or events not included in CTCAE were graded using tables provided in the study protocol.
Arm/Group | Tecovirimat | Placebo
All-Cause Mortality (participants affected / at risk) | 5/295 | 5/302
Serious Adverse Events (participants affected / at risk) | 15/295 | 15/302
Other Adverse Events (participants affected / at risk) | 214/295 | 211/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecovirimat (N=295) | Placebo (N=302)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Complicated malaria (Infections and infestations) | 2 (2) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Keratitis viral (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion early (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecovirimat (N=295) | Placebo (N=302)
Anaemia (Blood and lymphatic system disorders) | 16 (16) | 19 (19)
Abdominal pain (Gastrointestinal disorders) | 31 (32) | 26 (26)
Pyrexia (General disorders) | 39 (40) | 43 (47)
Malaria (Infections and infestations) | 34 (35) | 54 (55)
Haemoglobin decreased (Investigations) | 15 (15) | 18 (18)
Decreased appetite (Metabolism and nutrition disorders) | 20 (20) | 14 (14)
Headache (Nervous system disorders) | 20 (20) | 28 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 30 (32)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 27 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (15) | 18 (19)
Skin lesion (Skin and subcutaneous tissue disorders) | 13 (13) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT05559099/Prot_003.pdf
  • Statistical Analysis Plan: Main (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT05559099/SAP_004.pdf
  • Statistical Analysis Plan: Appendix 3 (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT05559099/SAP_005.pdf
  • Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT05559099/ICF_000.pdf